CLINICAL TRIAL: NCT06086197
Title: Prospective, Single-center, Phase II Clinical Study of Anlotinib in Combination With Rituximab，Gemcitabine and Oxaliplatin (A-RGEMOX) in the Treatment of Early Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: A-RGEMOX in the Treatment of Early Relapsed/Refractory DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A+RGEMOX
Record Dates: First submitted 2023-09-17; First posted 2023-10-17 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Diffuse Large B-cell Lymphoma Recurrent; Diffuse Large B Cell Lymphoma Refractory
Keywords: angiogenesis; anlotinib; early relapse; treatment
MeSH Terms: conditions — Recurrence | interventions — Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A+RGEMOX (Experimental): A-RGEMOX regimen (21 days per cycle, A total of 6 cycles) :
  Allotinib: 12mg d1~14 po qd, Rituximab: 375mg/m2 d1, gemcitabine: 1000mg/m2 d1 and d8, oxaliplatin: 130mg/m2 d1
  Interventions: Drug: Anlotinib hydrochloride, Rituximab, gemcitabine, oxaliplatin

INTERVENTIONS:
Drug: Anlotinib hydrochloride, Rituximab, gemcitabine, oxaliplatin — Anlotinib: 12mg d1~14 po qd, Rituximab: 375mg/m2 d1, gemcitabine: 1000mg/m2 d1 and d8, oxaliplatin: 130mg/m2 d1;
  For subjects ≥75 years of age, appropriate reduction of chemotherapy drugs (not less than 75% of the standard dose, or withdrawal of day 8 gemcitabine) may be decided by the investigator.

SUMMARY:
As the most common subtype of lymphoma, diffuse large B-cell lymphoma (DLBCL) is an aggressive but potentially curable malignancy. However, patients with early relapse (relapse within 12 months since diagnosis or the end of first-line treatment, ER) or primary refractory had an even worse prognosis. Thus, the investigators plan to evaluate the efficacy and safety of anlotinib combined with rituximab, gemcitabine, oxaliplatin (A-RGEMOX) in the treatment of early relapsed/refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL), the most common subtype of lymphoma, accounts for about 30%-40% of non-Hodgkin's lymphomas and is highly heterogeneous in terms of clinical presentation and biological behavior. About 10% of patients are resistant to first-line immunochemotherapy, and up to 30%-40% of patients will relapse after treatment. Patients with relapsed/refractory (R/R) DLBCL showed poor prognosis, with a median overall survival of only 6.3 months. Those with early relapse (relapse within 12 months since diagnosis or the end of first-line treatment, ER) or primary refractory had an even worse prognosis. So there is an unmet need for treatment in this population. Previous reports and our unpublished data showed the potential connection between angiogenesis and first-line treatment failure. Accordingly, we assume that the combination of anlotinib and RGEMOX regimen may improve the response rate of patients with early relapsed/refractory DLBCL, increasing the feasibility of follow-up ASCT, and improving long-term survival of this subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the clinical study voluntarily: fully understand and be informed of the study and sign the informed consent in person; Willing to follow and be able to complete all test procedures.
* Age≥18 years old, ECOG score ≥2 points, both male and female.
* Histopathologically confirmed as diffuse large B-cell lymphoma, not otherwise specified; high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement; high-grade B-cell lymphoma, not otherwise specified; EBV positive diffuse large B-cell lymphoma
* Must meet one of the following conditions:

  1. Early relapse: response (≥PR) to first-line systemic therapy (including rituximab and anthracyclines) and disease progression within 12 months after the end of treatment;
  2. Refractory: first-line treatment includes rituximab and anthracyclines, and no response has been achieved with the most recent systemic treatment (≥PR).
* At least one evaluable or measurable lesion that meets Lugano2014 criteria (evaluable lesion: PET/CT examination showing increased uptake in lymph nodes or extranodal areas (higher than liver) and PET/CT and/or CT consistent with lymphoma; Measurable lesions: nodular lesions >15mm in length or extragendal lesions >10mm in length with increased FDG uptake).
* Adequate organ and bone marrow function, no serious hematopoietic dysfunction, abnormal heart, lung, liver, kidney function and immune deficiency:

  1. Neutrophil absolute count (ANC) ≥1.5×109/L (1500/mm3), platelet ≥75×109/L, hemoglobin ≥100g/L (if bone marrow is involved, platelet ≥50×109/L, ANC ≥1.0×109/L, hemoglobin ≥80g/L).
  2. Liver function: serum bilirubin ≤2.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5 times the upper limit of normal value (AST or ALT≤5 times the upper limit of normal value is allowed if liver is involved).
  3. Renal function: creatinine clearance ≥60 mL/min (estimated according to the Cockcroft-Gault formula).
  4. Coagulation function: INR≤1.5 times the upper limit of normal value; PT and APTT≤1.5 times the upper limit of normal value.
* Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.
* Negative serum pregnancy test and effective contraceptive use from signing informed consent until 6 months after the last chemotherapy.
* Life expectancy > 3 months.

Exclusion Criteria:

* Pathological subtypes: primary central nervous system diffuse large B-cell lymphoma, primary mediastinal large B-cell lymphoma.
* Hemophagocytic syndrome at the time of diagnosis.
* Central nervous system involvement secondary to lymphoma.
* Participating in other clinical studies, or the first study drug is administered less than 4 weeks after the end of treatment in the previous clinical study.
* Medical history of other active malignancy within 2 years prior to enrollment, except for the following conditions:(1) adequately treated in situ of the cervix carcinoma; (2) local basal cell carcinoma or squamous cell carcinoma of skin; (3) Pre-existing malignant disease that is under control and has undergone local radical treatment (surgical or other forms).
* History of Human Immunodeficiency Virus (HIV) infection and/or acquired Immunodeficiency syndrome. Patients with positive hepatitis B surface antigen or hepatitis C virus antibody must be tested hepatitis B virus DNA (no more than 1000 iu/ml) and HCV RNA detection (below the detection limit). Patients with hepatitis B virus carriers, or stabilized hepatitis B with anti-virus treatment and cured hepatitis C can be included.
* Major surgery was performed within 28 days prior to study initiation.
* Any active infection, including bacterial, fungal or viral infections, that requires systemic antiinfection therapy within 14 days prior to treatment.
* Accompanied with severe or uncontrolled disease, including symptomatic of congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer or A history of severe hemorrhagic diseases, such as hemophilia A, hemophilia B, von willebrand disease or blood transfusion or other medical intervention history of spontaneous bleeding.
* History of stroke or intracranial hemorrhage within 6 months prior to first administration of the study drug.
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months.
* Patients who must take antiplatelet drugs and anticoagulants at the same time due to underlying diseases, and there is no alternative treatment plan.
* Continuous treatment with strong CYP1A2 and CYP3A inhibitors or inducers is required. Patients were excluded if they had taken a strong CYP1A2 and CYP3A inhibitors or inducer within 7 days prior to the first administration of the study drug (or had taken these drugs for less than 5 half-lives).
* Hypersensitivity to the experimental drug is known.
* Patients deemed unsuitable for the study by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CRR | 21days after the end of treatment
  Complete Remission Rate

SECONDARY OUTCOMES:
ORR | 21days after the end of treatment
  overall response rate
PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  Progression Free Survival
OS | From date of enrollment until the date of first documented date of death from any cause, assessed up to 5 years
  Overall Survival
PRR | 21days after the end of treatment
  Partial Remission Rate
AE and SAE | From date of first day of treatment until 30 day after last treatment
  Adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Yang, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No